CLINICAL TRIAL: NCT01770873
Title: Take Charge 2- A Multi-Center Randomized Trial of Mentoring to Prevent Youth Violence: Incorporating New Communication and Information Technology
Brief Title: A Multi-Center Randomized Controlled Trial of Mentoring to Prevent Youth Violence
Acronym: TC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NA_00075613; TC2-2P20 (Other: Other); 2P20MD000198-11 (NIH)
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Violence
Keywords: Youth; Violence; Assault-injured; Mentoring; Emergency Room; Urban
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Take Charge 2 (Experimental): Receipt of BBBS mentoring plus youth and parent violence prevention curriculum
  Interventions: Behavioral: Take Charge 2
- Control (No Intervention): Standard emergency room protocol followed

INTERVENTIONS:
Behavioral: Take Charge 2 — Youth assigned to the intervention receive a Big Brothers, Big Sisters (BBBS) mentor. During the match process, BBBS staff provide 3 session on violence prevention for the youth's parents. Six months into the mentoring relationship, mentors provide 6 sessions on violence prevention for the youth.
  Arms: Take Charge 2

SUMMARY:
The purpose of this study is to test whether a violence prevention curriculum delivered by Big Brothers and Big Sisters staff and mentors can reduce violence involvement for assault-injured youth.

DETAILED DESCRIPTION:
Violent injury is a major cause of morbidity and mortality among adolescents. The presence of a positive adult role model is a well-established protective factor against violence and other maladaptive outcomes among youth. Big Brothers Big Sisters (BBBS) is the largest U.S. mentoring organization with proven effectiveness in improving youth outcomes. However, these programs may be less effective with youth who already are exhibiting involvement in problem behavior at the time of program referral. Take Charge!, a mentor- and professional-implemented intervention with 10-15 year old assault-injured youth, showed promise for improving perceived self efficacy for avoiding violence and for decreasing aggression and problem behavior.

The overall goal of the proposed project is to develop, implement, and evaluate a research-informed youth development program that adapts the BBBS model to work for assault-injured youth. The aims are:

* To expand and refine Take Charge! and integrate it with BBBS practices;
* To conduct a randomized, controlled trial in which assault-injured 10-15 year old youth recruited from emergency departments in Baltimore and D.C. receive either standard emergency department follow-up care or the Take Charge! 2 intervention with assessment of violence-related, mental health, and educational outcomes;
* To conduct a comprehensive process evaluation of Take Charge! 2;
* And to accurately measure the costs of the intervention and assess cost-effectiveness.

Youth violence is a major cause of morbidity and mortality with marked disparities by race/ethnicity and socioeconomic status. This study is a critical next step in translating evidence-based research to real-world settings and practice.

ELIGIBILITY:
Inclusion Criteria:

* Treatment for an assault injury in the emergency room
* English speaking (parent and youth)

Exclusion Criteria:

* Treatment for child abuse, sexual abuse, sibling fights, or police fights
* Severe psychopathology

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2013-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Fighting | Past 30 days
  Have you been in a physical fight in the past 30 days?

CONTACTS AND LOCATIONS:
Overall Officials: Tina L Cheng, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Lindstrom Johnson S, Jones V, Ryan L, DuBois DL, Fein JA, Cheng TL. Investigating Effects of Mentoring for Youth with Assault Injuries: Results of a Randomized-Controlled Trial. Prev Sci. 2022 Nov;23(8):1414-1425. doi: 10.1007/s11121-022-01406-z. Epub 2022 Jul 25. PMID 35877056